CLINICAL TRIAL: NCT06599879
Title: Irradiation in Paediatrics: Neurocognition, Neuroimaging and Evaluation of Memory and Attention
Acronym: IPANEMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24TETE01
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor, Pediatric
Keywords: Brain Tumor, Pediatric; Radiotherapy; Neurocognitive sequelae; Imaging
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a brain tumour treated with radiotherapy in the first line 2 years prior to inclusion. (Other)
  Interventions: Other: Neuropsychological assessments:

INTERVENTIONS:
Other: Neuropsychological assessments: — Several neuropsychological assessments were carried out during the study (at inclusion and 2 years after inclusion), consisting of :
  * parental questionnaires (standard questionnaires and questionnaires specifically drawn up for the trial). The aim of these questionnaires will be to assess the patient's neurocognitive level at different times (before and after radiotherapy treatment).
  * patient cognitive tests (½ day face-to-face consultation/assessment with a neuropsychologist specialising in paediatrics, followed by a 30-minute telephone call).
  Only for patients having received their radiotherapy treatment at the IUCT-O: a multimodal MRI specific to the study (without injection of contrast product) may be performed at inclusion and 2 years after inclusion.

SUMMARY:
This is a prospective, open-label, multicentric study designed to correlate the dose delivered to the hippocampus with declarative memory deficits 2 years after radiotherapy treatment in a paediatric population who had received brain irradiation between the ages of 4 and 12 for a brain tumour.

In order to meet this objective, several neuropsychological assessments consisting of parental questionnaires and cognitive tests will be carried out during the course of the study, at the following two stages:

* A 1st assessment at patient inclusion, i.e. 2 years after the end of radiotherapy treatment,
* And a second assessment 2 years after patient inclusion, i.e. 4 years after the end of radiotherapy treatment.

A retrospective assessment of the patient's neurocognitive level 1 year before the diagnosis of the disease will also be carried out at inclusion, with the parents completing a questionnaire specifically designed for the trial.

In addition, patients who have received their radiotherapy treatment at the IUCT-O will be offered participation in the ancillary imaging study. If the parents and the patient agree, multimodal MRI scans specific to the study (without injection of contrast) will be performed at inclusion and 2 years after inclusion.

Imaging and radiotherapy data will be collected in parallel using the PediaRT software used in current practice (collection of radiotherapy dosimetric data as well as standard MRI examinations pre-operatively, post-operatively, and at the 2-year and 4-year follow-up).

130 patients will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who has received localised brain irradiation or craniospinal irradiation for a brain tumour whose treatment includes first-line radiotherapy.
2. Patient with one of the following tumour types: ependymomas, medulloblastomas, malignant germ cell tumours, craniopharyngioma, pinealoblastoma.
3. Patient aged between 4 and 12 years at the time of radiotherapy treatment.
4. End of irradiation within 2 years (+/-3 months) prior to inclusion.
5. Patient having been treated by photontherapy or proton therapy.
6. Sufficient visual, auditory (with authorised hearing aid) and oral or written expression capacity to carry out the neuropsychological tests properly.
7. Proficiency in the French language by the patient and parent(s).
8. Patient affiliated to a Social Security scheme in France.
9. Informed consent signed by the patient/legal parent(s)/guardian(s) in accordance with French law and Good Clinical Practice.

Exclusion Criteria:

1. Patient presenting with severe ataxia.
2. Patient with a recurrence of the disease.
3. Not applicable since protocol version 2. Metastatic patient.
4. Any contraindication to MRI for patients included in Toulouse (i.e. in particular patients with a pacemaker or cardiac defibrillator, implanted equipment activated by an electrical, magnetic or mechanical system, patients with haemostatic clips on intracerebral aneurysms, patients with orthopaedic implants, claustrophobic patients).
5. Patients undergoing psychostimulant or psychotropic treatment (in particular methylphenidate, antidepressants).
6. Any psychological, family, geographical or sociological condition that prevents compliance with medical monitoring and/or the procedures set out in the study protocol.
7. Patients deprived of their liberty or under legal protection.
8. Severe posterior fossa syndrome with akinetic mutism.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2030-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
A deficit of the declarative memory will be defined by a standard score of the Children' Memory Scale (CMS) ≤ 5 | 24 months for each patient

SECONDARY OUTCOMES:
Declarative memory will be assessed using the adapted EPIREAL test. | 24 months for each patient
Declarative memory will be assessed by the autobiographical memory question. | 24 months for each patient
The deficit of the procedural memory will be defined by a score of less than or equal to 10/20 on the last 20 trials (out of 50) of the probabilistic classification task. | 24 months for each patient
The deficit of the procedural memory will be defined by a specific learning score less than or equal to zero of the adapted serial reaction time task (SRTT). | 24 months for each patient
Working memory deficit will be defined if at least one of the two subtests (Number memory (WISC-V) and Spatial memory (WNV)) shows a deficit. | 24 months for each patient
  For each subtest, a deficit will be defined respectively by a standard score ≤ 5 and a percentile rank ≤ 5.

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - APHM - Hôpital la Timone, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - Institut Curie, Paris
  - Centre Eugène Marquis, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - IUCT-O, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif